CLINICAL TRIAL: NCT06384014
Title: Comparison of the Effect of Orthograde and Retrograde Mineral Trioxide Aggregate Application on Healing After Apical Resection in Teeth With Periapical Lesions
Brief Title: Examining the Effect of Different Filling Techniques on Healing in Lesional Teeth
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ipek Eraslan Akyuz, research assistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/56
Record Dates: First submitted 2024-04-18; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Apical Cyst
MeSH Terms: conditions — Radicular Cyst

STUDY DESIGN:
Intervention Model Description: İki farklı grupta farklı kanal dolum teknikleri uygulandıktan sonra apikal rezeksiyon yapılarak lezyon iyileşmesinin değerlendirilmesi
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Retrograde canal filling technique (Active Comparator): Apical resection application after retrograde root canal filling
  Interventions: Device: retrograde and orthograde root canal filling
- Orthograde canal filling technique (Active Comparator): Apical resection application after orthograde root canal filling
  Interventions: Device: retrograde and orthograde root canal filling

INTERVENTIONS:
Device: retrograde and orthograde root canal filling — Apical resection application after root canal filling

SUMMARY:
Microorganisms are an important factor in the development of periradicular diseases. The goal of non-surgical endodontic treatment is to eliminate microorganisms and their byproducts from the root canal system and to create an effective barrier between the root canal system and surrounding tissues. If there is no healing in the periradicular tissues after non-surgical endodontic treatment or if retreatment becomes impossible, surgical endodontic treatment is required. Apical resection is a surgical technique that involves removing the root tip of the tooth and closing the apical portion of the root canal system. An ideal retrograde filling material should be non-toxic, non-carcinogenic and biocompatible. It must also have dimensional stability and sealing properties. Amalgam, glass ionomer cements, and zinc oxide-eugenol based materials have been used for root end fillings in periapical surgery, but the desired success was not achieved. Today, Mineral Trioxide Aggregate (MTA) is preferred as a retrograde filling material due to its superior sealing properties, ability to harden in the presence of blood and moisture, antibacterial effects, biocompatibility and radiopacity.

In the researchers' study, the effect of apical resection after orthograde canal filling and retrograde canal filling during apical resection on postoperative recovery will be compared. In both canal filling techniques, Sure-Seal Root MTA (Sure Dent Corporation-Korea) will be used as the filling material. Sure-Seal Root MTA is a calcium silicate based paste that is typically pre-mixed and ready to apply, exhibits excellent physical properties and does not show shrinkage during the curing process. As the manufacturer states, it is hydrophilic, biocompatible, has ideal setting and working time.

Our faculty has piezosurgical ultrasonics (Mectron ®, Grassobbio BG, Italy). After the root tip resection is performed, the retrograde cavity will be prepared with Woodpecker ultrasonic tips (Guilin, China) compatible with this device. In our study using these materials and devices, a comparative analysis of the effects of different canal filling techniques on lesion healing and improvement in clinical symptoms will be made.

DETAILED DESCRIPTION:
Periapical or periradicular lesions are barriers that restrict microorganisms and prevent their spread to surrounding tissues; microorganisms cause periapical lesions, either primary or secondary. Apical infections, if left untreated, can follow two different paths: First, the infection can create a path inside or outside the mouth, causing the pus to drain out. Secondly, infection within the canal; It may reach the periapical tissues and create a cavity surrounded by polymorphonuclear leukocytes in the bone, leading to the formation of inflammatory radicular cysts.

Inflammatory radicular cysts (IRCs) are chronic lesions that occur after the development of periapical granulomas (PGs). PGs and IRCs are thought to follow pulp infections as an inflammatory process at the periapical level. Although both conditions, PG and IRC, are clinically diagnosed as apical periodontitis (AP), they differ significantly histopathologically.

The majority of apical cysts are asymptomatic and may develop insidiously by being discovered incidentally during a routine x-ray examination as a large periapical radiolucency covering the apex of one or more teeth. By confirming that the lesion is a granuloma or cyst, a more definitive diagnosis is reached by histopathological examination. Although conventional radiographic methods cannot be used for the definitive diagnosis of periapical cysts, larger round or oval, well-circumscribed radiolucent images around the apex of the tooth are considered to be cystic lesions.

When the infection in the canal is successfully treated, apical cysts can regress by the apoptosis mechanism in the root canal without the need for surgical intervention. Researchers stated that incorrect histopathological diagnosis in early studies created the false impression that radicular cysts were more common, and that this methodological error led to the illusion that most cystic lesions in the periapex area healed after non-surgical root canal treatment. In conclusion, the authors suggested that true cysts may be less likely to heal with nonsurgical root canal treatment due to their inherently self-sustaining properties and may require surgical intervention. Whether true cysts heal after non-surgical root canal treatment is still a major debate.

Different retrograde canal filling materials have been tried in the literature, but today, Mineral Trioxide Aggregate (MTA) is most commonly used because it is more biocompatible and has a periapical healing-inducing effect. MTA; It is the first restorative material that allows cementum development and provides regeneration in periodontal ligament cells. In addition, histological sections taken from the periapical region of teeth with retrograde canal filling with MTA often showed new cementum formation not only on the resection surface but also directly on the MTA. For this reason, MTA is called bioactive material. Properties of MTA such as biocompatibility, sealing, and the capacity to increase the regeneration of pulp and periradicular tissues; It has increased the diversity of dental usage areas and clinical success rates, and has become the focus of attention of clinicians with this innovative structure. In comparative studies on retrograde filling materials, MTA has demonstrated an excellent tissue response with almost no inflammatory component.

There are few studies in the literature comparing the effects of two different canal filling techniques (orthograde, retrograde), which are currently frequently used, on postoperative recovery. There is no study comparing the long-term postoperative radiographic and clinical improvement levels of using MTA with different application techniques in teeth with periapical lesions with an indication for apical resection. The purpose of researchers' planned study is to compare and evaluate the healing effect of orthograde MTA application followed by resection in teeth with large periapical lesions and retrograde MTA application during apical resection operation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers without systemic disease between the ages of 18 and 65
* Single-rooted teeth with periapical lesions larger than 1 cm
* Patients who do not have any contraindications for the surgical procedure.

Exclusion Criteria:

* Individuals with systemic diseases and allergic reactions
* Pregnancy and breastfeeding
* Severely damaged teeth
* Patients with contraindications for surgical operation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of lesion healing rate after apical resection using different root canal filling techniques | 2 years
  lesion healing rate

CONTACTS AND LOCATIONS:
Overall Officials: ERASLAN AKYÜZ, Principal Investigator — BAŞ ARAŞTIRMACI; TOPÇUOĞLU, Study Director — YÜRÜTÜCÜ; ÖZDEMİR, Study Chair — YARDIMCI ARAŞTIRMACI
Locations (1):
- Erciyes Üniversitesi Diş Hekimliği Fakültesi, Kayseri, Turkey (Türkiye)